CLINICAL TRIAL: NCT03006328
Title: Technology-Assisted Weight Management Intervention Within Patient-Centered Medical Homes: The GEM (Goals for Eating and Moving) Study
Brief Title: The GEM (Goals for Eating and Moving) Study
Acronym: GEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-01445
Record Dates: First submitted 2016-12-20; First posted 2016-12-30 (Estimated); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Weight Gain; Obesity
Keywords: weight gain; weight loss
MeSH Terms: conditions — Weight Gain; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with Obesity + GEM (Experimental): Body mass index of ≥30kg/m2 OR Body mass index of ≥25 kg/m2 with an obesity associated co-morbidity. Will be assigned to GEM Tool and a health coach.
  Interventions: Behavioral: GEM
- Participants with Obesity + Enhanced Usual Care (Active Comparator): Body mass index of ≥30kg/m2 OR Body mass index of ≥25 kg/m2 with an obesity associated co-morbidity. Will receive receive non-tailored weight management handouts by health coaches.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: GEM — Online program designed to support health coach and primary care team counseling. It assesses current behaviors, barriers, and facilitators to weight loss via a 16-item questionnaire, provides tailored advice, and guides patients to set weight loss (5-10%), diet, and physical activity (PA) goals. After completing the tool, participants will meet with a Health Coach. Participants will receive 12 telephone coaching calls by a health coach over 12 months.
  Arms: Participants with Obesity + GEM
Behavioral: Enhanced Usual Care — Patients in the EUC arm will receive non-tailored weight management handouts. Patients will follow-up with their primary care teams as needed.
  Arms: Participants with Obesity + Enhanced Usual Care

SUMMARY:
The GEM intervention leverages the patient-centered medical home model by using the GEM tool to provide individually tailored, patient-centered care, promote standardized weight management counseling by health coaches and primary team members, coordinate care between teams and other weight management service providers/programs (e.g., dietitians, health educators, DPP), and provide feedback to the provider and primary care team about patients' weight management-related goals, progress, and care.

DETAILED DESCRIPTION:
To establish the efficacy of the GEM intervention, investigators will conduct a cluster randomized controlled 12-month intervention of 19 primary care teams at two urban healthcare systems with Medical Home models of care to compare the GEM intervention (intervention arm) with Enhanced Usual Care (educational materials; control arm).

The specific aims of this study are:

* Test the impact of the GEM intervention on weight change, and clinical and behavioral outcomes.
* Identify predictors of weight loss in the GEM intervention arm related to: a) goal-setting processes and b) intervention components
* Determine the impact of the GEM intervention on obesity-related counseling practices and attitudes in primary care providers.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-69 years of age,
* Body mass index of ≥30kg/m2 OR
* Body mass index of ≥25 kg/m2 with an obesity associated co-morbidity
* Hypertension
* High Cholesterol
* Sleep Apnea
* Osteoarthritis
* Metabolic Syndrome
* Prediabetes
* Under primary care team care with at least one prior visit with their provider in the past 24 months
* Access to a telephone, and ability to travel for in-person evaluations at baseline, 6, 12, and 24 months

Exclusion Criteria:

* Patients who do not speak English or Spanish,
* Have active psychosis or other cognitive issues,
* Psychoactive substance use
* Diabetes
* Taking prescription weight-loss medication
* Health condition that may prohibit the patient from walking or physical activity such as chest tightness, a heart condition, or severe arthritis
* Participated in MOVE!, DPP, or another intensive weight management program (>3 sessions) in the past year,
* Have a history of bariatric surgery,
* Are pregnant, or become pregnant during the intervention period,
* Metastatic cancer in the last 6 months, current chemotherapy or cancer treatment,
* Have a provider who states they should not participate,
* Patients who do not want to lose weight
* Have self-reported inability to read at 5th grade level.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Jay, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University Medical Center Institutional Review Boards, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Merriwether EN, Wittleder S, Cho G, Bogan E, Thomas R, Bostwick N, Wang B, Ravenell J, Jay M. Racial and weight discrimination associations with pain intensity and pain interference in an ethnically diverse sample of adults with obesity: a baseline analysis of the clustered randomized-controlled clinical trial the goals for eating and moving (GEM) study. BMC Public Health. 2021 Dec 2;21(1):2201. doi: 10.1186/s12889-021-12199-1. PMID 34856961
- [Derived] Wittleder S, Ajenikoko A, Bouwman D, Fang Y, McKee MD, Meissner P, Orstad SL, Rehm CD, Sherman SE, Smith S, Sweat V, Velastegui L, Wylie-Rosett J, Jay M. Protocol for a cluster-randomized controlled trial of a technology-assisted health coaching intervention for weight management in primary care: The GEM (goals for eating and moving) study. Contemp Clin Trials. 2019 Aug;83:37-45. doi: 10.1016/j.cct.2019.06.005. Epub 2019 Jun 20. PMID 31229622
- [Derived] Viglione C, Bouwman D, Rahman N, Fang Y, Beasley JM, Sherman S, Pi-Sunyer X, Wylie-Rosett J, Tenner C, Jay M. A technology-assisted health coaching intervention vs. enhanced usual care for Primary Care-Based Obesity Treatment: a randomized controlled trial. BMC Obes. 2019 Feb 4;6:4. doi: 10.1186/s40608-018-0226-0. eCollection 2019. PMID 30766686

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Care Clusters
Period: Overall Study
Arm/Group | Participants With Obesity + GEM | Participants With Obesity + Enhanced Usual Care
Started | 220; 9 Care Clusters | 269; 10 Care Clusters
Completed | 220; 9 Care Clusters | 269; 10 Care Clusters
Not Completed | 0; 0 Care Clusters | 0; 0 Care Clusters

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Obesity + GEM | Participants With Obesity + Enhanced Usual Care | Total
Number analyzed (Participants) | 220 | 269 | 489
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.1) | 50.2 (11.6) | 49.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 157 | 273
  Male | 104 | 112 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 99 | 100 | 199
  Not Hispanic or Latino | 116 | 166 | 282
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 96 | 142 | 238
  White | 35 | 41 | 76
  More than one race | 6 | 10 | 16
  Unknown or Not Reported | 80 | 72 | 152
Region of Enrollment [Number; unit: participants]
  United States | 220 | 269 | 489

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Participants With Obesity + GEM | Participants With Obesity + Enhanced Usual Care
Number analyzed (Participants) | 220 | 269
kilograms | -1.4 (0.8) | -0.8 (0.9)

2. Primary Outcome: Change in Waist Circumference From Baseline
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Participants With Obesity + GEM | Participants With Obesity + Enhanced Usual Care
Number analyzed (Participants) | 220 | 269
centimeters | -1.3 (0.5) | -0.6 (0.6)

3. Primary Outcome: Change in Systolic Blood Pressure (SBP) From Baseline
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Participants With Obesity + GEM | Participants With Obesity + Enhanced Usual Care
Number analyzed (Participants) | 220 | 269
mmHg | 1.8 (1.7) | 3.2 (1.7)

4. Primary Outcome: Change in Diastolic Blood Pressure (DBP) From Baseline
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Participants With Obesity + GEM | Participants With Obesity + Enhanced Usual Care
Number analyzed (Participants) | 220 | 269
mmHg | 1.6 (1.4) | 3.2 (1.5)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Participants With Obesity + GEM | Participants With Obesity + Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 1/220 | 3/269
Serious Adverse Events (participants affected / at risk) | 53/220 | 81/269
Other Adverse Events (participants affected / at risk) | 36/220 | 43/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Obesity + GEM (N=220) | Participants With Obesity + Enhanced Usual Care (N=269)
Depression (Psychiatric disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal Surgery (Surgical and medical procedures) | 4 | 0
Gallbladder Disease (Gastrointestinal disorders) | 0 | 4
Allergic Reaction (Immune system disorders) | 0 | 2
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Appendix Removed (Surgical and medical procedures) | 1 | 0
Possible Panic Attack (Psychiatric disorders) | 1 | 0
Scrotal Pain (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Autoimmune Disorder on Eye (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Sepsis (Infections and infestations) | 1 | 0
Biopsy resulted in needing catheterization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blood Transfusion (Blood and lymphatic system disorders) | 0 | 2
hypertension (Vascular disorders) | 2 | 0
Breast Cancer Surgery (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leg fracture (Injury, poisoning and procedural complications) | 1 | 0
Motor vehicle accident (Injury, poisoning and procedural complications) | 3 | 3
Cardiac heart catheterization (Cardiac disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 4 | 1
Complications after biopsy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Severe pain in feet (Musculoskeletal and connective tissue disorders) | 0 | 1
COVID-19 infection (Infections and infestations) | 1 | 1
Wound requiring stitches (Injury, poisoning and procedural complications) | 0 | 1
Diverticulitis (Gastrointestinal disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 2 | 5
Gout (Musculoskeletal and connective tissue disorders) | 0 | 2
Upper Respiratory Infection (Infections and infestations) | 1 | 2
Heart and blood vessel issues (Cardiac disorders) | 0 | 1
Heart Attack (Cardiac disorders) | 1 | 0
Hemorrhage (Blood and lymphatic system disorders) | 0 | 1
Hernia (Musculoskeletal and connective tissue disorders) | 1 | 0
Severe muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Arm paralysis secondary to botox injection (Injury, poisoning and procedural complications) | 1 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Kidney pain/stones (Renal and urinary disorders) | 2 | 3
Knee pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Knee surgery (Surgical and medical procedures) | 1 | 1
Lumbar scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metal in eye, work injury (Injury, poisoning and procedural complications) | 0 | 1
Migraines (Nervous system disorders) | 0 | 2
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Loss of consciousness/fainting (Nervous system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Wrist/hand injury (Injury, poisoning and procedural complications) | 0 | 5
Upper respiratory infection (Infections and infestations) | 0 | 1
Prostate Cancer Operation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Retina Surgery (Eye disorders) | 0 | 2
Seizure (Nervous system disorders) | 0 | 1
Skin cancer removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small tumor found on kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal operation (Surgical and medical procedures) | 1 | 2
Cardiac Arrythmia (Cardiac disorders) | 0 | 2
Stroke (Nervous system disorders) | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Surgery for parathyroid removal (Surgical and medical procedures) | 0 | 1
Broken ribs (Injury, poisoning and procedural complications) | 1 | 0
Urology surgery (Surgical and medical procedures) | 0 | 1
Vertigo (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Work accident (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Obesity + GEM (N=220) | Participants With Obesity + Enhanced Usual Care (N=269)
Depression (Psychiatric disorders) | 2 | 0
Abcess (Skin and subcutaneous tissue disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Acute muscle spasm (Musculoskeletal and connective tissue disorders) | 2 | 0
Allergic reaction (Immune system disorders) | 1 | 1
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 | 0
Catheter Adjusted Due to Discomfort (Surgical and medical procedures) | 0 | 1
Catheter Removed (Surgical and medical procedures) | 0 | 1
Victim of assault (Injury, poisoning and procedural complications) | 0 | 1
Chest pains (Cardiac disorders) | 5 | 0
Headaches from sinus issues (General disorders) | 0 | 1
COVID-19 infection (Infections and infestations) | 0 | 4
Cyst in arm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Endoscopy and colonoscopy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Enlarged Prostate (Reproductive system and breast disorders) | 0 | 1
Plantar faciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Upper Respiratory Infection (Infections and infestations) | 1 | 2
Wrist/hand injury (Injury, poisoning and procedural complications) | 2 | 3
Kidney pain/stones (Renal and urinary disorders) | 0 | 1
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Lightheaded, dizzy (Nervous system disorders) | 1 | 0
Lipoma in left abdomen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Migraines (Nervous system disorders) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Ankle pain due to injury (Injury, poisoning and procedural complications) | 1 | 0
Injury requiring physical therapy (Injury, poisoning and procedural complications) | 1 | 0
Diffuse muscle pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fever (Infections and infestations) | 1 | 0
Shoulder pain/injury (Musculoskeletal and connective tissue disorders) | 3 | 5
Sinus infection (Infections and infestations) | 0 | 1
Sore throat (Infections and infestations) | 1 | 0
Staphylococcus aureus infection in leg (Infections and infestations) | 1 | 0
Tonsil Removal (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Foot sprain (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT03006328/Prot_SAP_000.pdf